CLINICAL TRIAL: NCT06461195
Title: Computer Aided Respiratory Therapy Based on Audio and Spirometry Signals
Acronym: COMPASS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lieven De Maesschalck (Other)
Collaborators: KU Leuven (Other); Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor-Investigator, Lieven De Maesschalck, Innovation Manager, Thomas More Kempen
Organization: Thomas More Kempen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023COMPASS-ST01
Record Dates: First submitted 2024-04-19; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Respiratory Therapy
Keywords: Spirometry; Respiratory sounds
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Intervention Model Description: Single group interventional study acquiring spirometry data, respiration sound and physiological data in patients suffering from pulmonary disease.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regular respiratory physiotherapy while being monitored (Experimental): Patients receive their standard respiratory physiotherapy, but in the mean time they are monitored with a stethoscope, spirometer and a wearable to measure physiological parameters.
  Interventions: Other: Monitoring of patients

INTERVENTIONS:
Other: Monitoring of patients — Data from a spirometer and a stethoscope are captured to develop algorithms to detect and classify respiration sounds to support therapists and patients in future therapy.

SUMMARY:
The purpose of the study is to collect data: audio in the form of respiratory sounds and instructions from the therapist, spirometry data during the execution of the therapy, physiological parameters, and patient information. With the help of this data, algorithms will be developed for the automatic detection, localization, and classification of respiratory sounds, linked to the respiratory cycle using spirometric signals.

DETAILED DESCRIPTION:
The study is an interventional study. Patients receive their standard respiratory physiotherapy, but in the mean time they are monitored with a stethoscope, spirometer and a wearable to measure physio-logical parameters.

It has been chosen to intervene as little as possible in the therapy to measure the respiratory sounds and breathing of the patient as accurately as possible. By recording therapy sessions with 15 patients, we expect to register several hundred events of respiratory sounds. This provides a good foundation for training an algorithm to detect and classify respiratory sounds.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a chronic or acute respiratory condition and may need oxygen therapy
* The patient is minimally 12 years old

Exclusion Criteria:

* The patient is cognitively impaired.
* The patient has an undrained pneumothorax.
* The patient is experiencing an acute pulmonary hemorrhage.
* The patient is having an asthma exacerbation.
* The patient has an infection with Burkholderia cepatia.
* The patient is in isolation due to the risk of infection.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-06-25 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Respiration flow | 1 year
  Measured in liter per minute, measured by a spirometer.
Respiration volume | 1 year
  Measured in liter, measured by a spirometer.

SECONDARY OUTCOMES:
Heart rate | 1 year
  Measured in beats per minute by photoplethysmography using a wrist watch with a sensor
Skin conductivity | 1 year
  Measured in Siemens using a wrist watch with a sensor
Body temperature | 1 year
  Measured in degrees Celsius using a wrist watch with a sensor
Oxygen saturation | 1 year
  Measured in percentage by photoplethysmography using a wrist watch with a sensor

CONTACTS AND LOCATIONS:
Overall Officials: Filip Van Ginderdeuren, PhD, Principal Investigator — Universitair Ziekenhuis Brussel

IPD SHARING:
Plan to Share IPD: No